CLINICAL TRIAL: NCT01382212
Title: A Phase 3, Open-Label, Multicenter Study to Evaluate the Safety of Paricalcitol Capsules in Pediatric Subjects Ages 10 to 16 With Stage 5 Chronic Kidney Disease Receiving Peritoneal Dialysis or Hemodialysis
Brief Title: A Study to Evaluate the Safety of Paricalcitol Capsules in Pediatric Subjects Ages 10 to 16 With Stage 5 Chronic Kidney Disease Receiving Peritoneal Dialysis or Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11-612; 2013-002610-13 (EudraCT Number)
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2016-11

CONDITIONS: End-Stage Renal Disease; Secondary Hyperparathyroidism
Keywords: Evaluate safety through the evaluation of the incidence of hypercalcemia in pediatric subjects
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperparathyroidism, Secondary | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paricalcitol (Experimental): Open-label paricalcitol (maximum dose of 16 µg), 3 times weekly (no more frequently than every other day) for 12 weeks.
  Interventions: Drug: paricalcitol

INTERVENTIONS:
Drug: paricalcitol — Paricalcitol soft capsule. Starting dose of paricalcitol was determined by the intact parathyroid hormone (iPTH) value (iPTH/120) from prior to Day 1, rounded down to the nearest whole number, not to exceed 16 µg 3 times weekly, no more frequently than every other day. Decisions to hold, maintain, increase, or decrease a dose were based on the iPTH, phosphorus, and calcium results generated from the most recent visit and within target Kidney Dialysis Outcomes Quality Initiatives (KDOQI) levels.
  Other Names: ABT-358, Zemplar

SUMMARY:
The objective is to evaluate the safety of paricalcitol capsules in pediatric subjects, ages 10 to 16 years old, with Stage 5 chronic kidney disease (kidney failure) receiving peritoneal dialysis or hemodialysis and being treated for secondary hyperparathyroidism. Subjects will be in the dosing period of the study for 12 weeks in order to evaluate the incidence of hypercalcemia (high calcium levels in blood). Approximately 12 subjects will be enrolled and all 12 will receive paricalcitol capsules.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be receiving peritoneal dialysis or hemodialysis for at least 3 months prior to Screening
* Subject is currently being diagnosed and/or treated for secondary hyperparathyroidism
* For entry into the Dosing Period (for subjects that are naïve to Vitamin D Receptor [VDR] Activators or those who have completed a 2 to 12 week washout), the subject must meet the following laboratory criteria prior to enrollment:

  * A corrected calcium value ≥ 8.2 and ≤ 10.4 mg/dL
  * A phosphorus value ≤ 6.5 mg/dL
  * An intact parathyroid hormone (iPTH) value > 300 pg/mL and less ≤ 2000 pg/mL

Exclusion Criteria:

* Subject is expected or scheduled to receive a living donor kidney transplant within 3 months of Screening or is a kidney transplant patient requiring full immunosuppressant therapy
* Subject is expected to stop peritoneal dialysis or hemodialysis within 4 months of Screening (per investigator discretion)
* Subject has had a parathyroidectomy within 12 weeks prior to Screening
* Subject has had symptomatic or significant hypocalcemia requiring VDR Activator therapy (i.e., calcitriol, paricalcitol, or doxercalciferol) within 2 months prior to Screening
* Subject is taking maintenance calcitonin, bisphosphonates, glucocorticoids in an equivalent dose of greater than 5 mg prednisone daily, or other drugs known to affect calcium or bone metabolism within 4 to 8 weeks prior to Dosing
* Subject is receiving cinacalcet at the time of Screening

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Eldred, MD, Study Director — AbbVie

REFERENCES:
- [Result] Webb NJA, Lerner G, Warady BA, Dell KM, Greenbaum LA, Ariceta G, Hoppe B, Linde P, Lee HJ, Eldred A, Dufek MB. Efficacy and safety of paricalcitol in children with stages 3 to 5 chronic kidney disease. Pediatr Nephrol. 2017 Jul;32(7):1221-1232. doi: 10.1007/s00467-017-3579-6. Epub 2017 Mar 22. PMID 28332096
- See also: Prescribing Information — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 26 subjects were screened and 13 pediatric subjects (between 10 and 16 years of age) were enrolled; 1 subject was 16 years of age at the time of Screening and turned 17 by the time treatment began.
Period: Overall Study
Arm/Group | Paricalcitol
Started | 13
Completed | 11
Not Completed | 2
Not completed — Kidney transplant | 1
Not completed — Withdrew consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Hypercalcemia
Description: The percentage of subjects with hypercalcemia, defined as at least 2 consecutive post-baseline corrected calcium values > 10.2 mg/dL (2.55 mmol/L).
Time Frame: Day 1 to Week 12
Population: All-treated data set: all subjects enrolled and administered at least 1 dose of paricalcitol
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
percentage of participants | 15.3 [1.9 to 45.4]

2. Secondary Outcome: Percentage of Subjects With 2 Consecutive Intact Parathyroid Hormone (iPTH)/120 Between 150 and 300 pg/mL
Time Frame: Baseline (last measurement collected prior to the first dose) to Week 12
Population: All-treated data set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
percentage of participants | 38.5 [13.9 to 68.4]

3. Secondary Outcome: Percentage of Subjects With 2 Consecutive iPTH Reductions of at Least 30% From Baseline
Time Frame: Baseline (last measurement collected prior to the first dose) to Week 12
Population: All-treated data set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
percentage of participants | 61.5 [31.6 to 86.1]

4. Secondary Outcome: Hemoglobin: Mean Change From Baseline to Final Visit
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 11
g/dL | -0.1 (1.263)

5. Secondary Outcome: Hematocrit: Mean Change From Baseline to Final Visit
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Paricalcitol
Number analyzed (Participants) | 11
percent | -1.08 (5.066)

6. Secondary Outcome: Red Blood Cells: Mean Change From Baseline to Final Visit
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: cells x 10^6/µL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 11
cells x 10^6/µL | -0.09 (0.496)

7. Secondary Outcome: White Blood Cells (WBC) and Platelet Count: Mean Change From Baseline to Final Visit
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: cells x 10^3/µL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 11
cells x 10^3/µL
  WBC | -0.06 (2.982)
  Platelet Count | 19.2 (47.03)

8. Secondary Outcome: Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils: Mean Change From Baseline to Final Visit
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: cells x 10^9/µL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 11
cells x 10^9/µL
  Neutrophils | 0.11 (2.6812)
  Lymphocytes | -0.294 (0.597)
  Monocytes | 0.032 (0.1276)
  Eosinophils | 0.059 (0.1522)
  Basophils | -0.01 (0.0322)

9. Secondary Outcome: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Lactic Dehydrogenase (LDH), and Bone-Specific Alkaline Phosphatase (BSAP): Mean Change From Baseline to Final Visit
Description: n=subjects with evaluable Baseline and Post-baseline data for each parameter.
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Paricalcitol
Number analyzed (Participants) | 11
U/L
  ALT (n=11) | -4.55 (16.501)
  AST (n=11) | -4.45 (12.25)
  LDH (n=11) | -6.5 (33.22)
  BSAP (n=9) | -49.4 (86.95)

10. Secondary Outcome: Bilirubin, Blood Urea Nitrogen (BUN), Uric Acid, Magnesium, Glucose, Cholesterol, Triglycerides, High Sensitivity C-Reactive Protein (hsCRP), Inorganic Phosphate, Corrected Calcium, and Creatinine: Mean Change From Baseline to Final Visit
Description: n=subjects with evaluable Baseline and Post-baseline data for each parameter.
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 11
mg/dL
  Total bilirubin (n=11) | 0.032 (0.3165)
  Direct Bilirubin (n=11) | 0.013 (0.0785)
  Indirect Bilirubin (n=9) | 0.056 (0.3035)
  BUN (n=11) | 1.33 (11.614)
  Uric Acid (n=11) | 0.31 (1.245)
  Magnesium (n=11) | 0.082 (0.3649)
  Glucose (n=11) | 4.36 (10.172)
  Cholesterol (n=11) | -16.4 (27.37)
  Triglycerides (n=11) | 9.2 (40.32)
  hsCRP (n=11) | 0.061 (0.1967)
  Inorganic phosphate (n=13) | 0.64 (1.188)
  Corrected Calcium (n=7) | 0.31 (0.421)
  Creatinine (n=11) | 0.48 (1.592)

11. Secondary Outcome: Alkaline Phosphatase: Mean Change From Baseline to Final Visit
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Paricalcitol
Number analyzed (Participants) | 11
IU/L | -61.8 (117.34)

12. Secondary Outcome: Sodium, Potassium, Chloride, Bicarbonate: Mean Change From Baseline to Final Visit
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Paricalcitol
Number analyzed (Participants) | 11
mEq/L
  Sodium | -0.5 (2.02)
  Potassium | 0.25 (0.746)
  Chloride | 0.5 (3.21)
  Bicarbonate | -0.45 (3.446)

13. Secondary Outcome: Total Protein and Albumin: Mean Change From Baseline to Final Visit
Description: n=subjects with evaluable Baseline and Post-baseline data for each parameter.
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All-treated data set
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
g/dL
  Total protein (n=11) | 0.15 (0.43)
  Albumin (n=13) | 0.04 (0.325)

14. Secondary Outcome: Fibroblast Growth Factor-23 (FGF-23), 1,25-Hydroxy Vitamin D, 25-Hydroxy Vitamin D, and Intact Parathyroid Hormone (iPTH): Mean Change From Baseline to Final Visit
Description: n=subjects with evaluable Baseline and Post-baseline data for each parameter.
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All-treated data set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
pg/mL
  FGF-23 (n=10) | 1990.7 (3317.7)
  1,25-Hydroxy Vitamin D (n=11) | 15.65 (29.296)
  25-Hydroxy Vitamin D (n=11) | 5.8 (10.38)
  iPTH (n=13) | -437.5 (491.83)

15. Secondary Outcome: Osteocalcin: Mean Change From Baseline to Final Visit
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All subjects in the all-treated data set with evaluable data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paricalcitol
Number analyzed (Participants) | 10
ng/mL | 117.21 (223.07)

16. Secondary Outcome: Number of Subjects With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug. For more details on adverse events please see the Adverse Event section.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to 16 weeks).
Population: All-treated data set
Measure: Number; unit: participants
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
participants
  Any TEAE | 11
  TESAE | 2

17. Secondary Outcome: Number of Subjects With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were recorded after the subject had been in the supine position for at least 5 minutes. The number of subjects with potentially clinically significant ECG findings, as determined by the investigator, is presented.
Time Frame: Baseline (Day 1) to Final Visit (up to Week 12)
Population: All-treated data set
Measure: Number; unit: participants
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
participants | 0

18. Secondary Outcome: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP): Mean Change From Baseline to Final Visit
Description: Blood pressure was measured after the subject had been sitting for at least 3 minutes.
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All-treated data set
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
mm Hg
  SBP | 7.5 (15.66)
  DBP | 3.7 (12.98)

19. Secondary Outcome: Heart Rate: Mean Change From Baseline to Final Visit
Description: Heart rate was measured after the subject had been sitting for at least 3 minutes.
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All-treated data set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
bpm | 1.8 (17.43)

20. Secondary Outcome: Oral Body Temperature: Mean Change From Baseline to Final Visit
Time Frame: Baseline (last measurement collected prior to the first dose) to Final Visit (up to Week 12)
Population: All-treated data set
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
degrees Celsius | 0.03 (0.338)

21. Secondary Outcome: Number of Subjects With Potentially Clinically Significant Physical Examination Findings
Time Frame: Baseline (Day 1) and Final Visit (up to Week 12)
Population: All-treated data set
Measure: Number; unit: participants
Arm/Group | Paricalcitol
Number analyzed (Participants) | 13
participants | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from first dose of study drug until 30 days following last dose of study drug (up to 16 weeks); serious adverse events were collected from the time when informed consent was obtained (up to 28 weeks).
Groups:
- Paricalcitol: Open-label paricalcitol (maximum dose of 16 μg), 3 times weekly (no more frequently than every other day) for 12 weeks.
Arm/Group | Paricalcitol
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=13)
PERITONEAL DIALYSIS COMPLICATION (Injury, poisoning and procedural complications) | 1
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=13)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 1
INFLUENZA LIKE ILLNESS (General disorders) | 1
PYREXIA (General disorders) | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1
PROCEDURAL VOMITING (Injury, poisoning and procedural complications) | 1
BLOOD CALCIUM INCREASED (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 1
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
HEADACHE (Nervous system disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 2
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
HYPERTENSION (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The sample size of the study was limited to 13 subjects and there was no comparator group, so the study was not designed to analyze efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.